CLINICAL TRIAL: NCT02316717
Title: A Phase ll, Randomized, Double-blind, Placebo-controlled Study of IMM-124E for Patients With Non-alcoholic Steatohepatitis.
Brief Title: A Phase ll Study of IMM-124E for Patients With Non-alcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immuron Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMM-124E-2001
Record Dates: First submitted 2014-11-06; First posted 2014-12-15 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-01

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Arm A (Experimental): IMM-124E, 600 mg three times daily, orally plus matching placebo
  Interventions: Biological: IMM-124E
- Treatment Arm B (Experimental): IMM-124E, 1200 mg three times daily, orally
  Interventions: Biological: IMM-124E
- Treatment Arm C (Placebo Comparator): Matching placebo, three times daily, orally
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IMM-124E — IMM-124E
  Arms: Treatment Arm A; Treatment Arm B
Other: Placebo — Matched placebo
  Arms: Treatment Arm C

SUMMARY:
This study will evaluate the safety and preliminary efficacy of two dose levels of IMM-124E in reducing liver fat and/or serum alanine aminotransaminase (ALT) compared with placebo.

DETAILED DESCRIPTION:
Subjects who provide voluntary written informed consent will be screened for eligibility. Subjects meeting all of the inclusion and none of the exclusion criteria will be eligible to participate.

Eligible subjects will be randomized at the Baseline visit to receive one of the three study treatments three times daily for a period of 24 weeks. Each subject will return to the study clinic for assessment and required study procedures on Day 7, 14 and 28 and every 4 weeks thereafter until Week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Provision of written informed consent.
3. Diagnosis of NASH, histologically proven within 12 months of Screening with

   * NASH activity score (NAS) of 4 or more
   * cytologic ballooning score of at least 1;
   * 10% or more macrovescicular steatosis.
   * Hematoxylin & Eosin (H&E) stained slides and/or paraffin block available for independent assessment.
4. HBA1C of <9.0
5. Agree to the use of effective contraceptive measures if either male or female of child bearing potential.

Exclusion Criteria:

1. Presence of vascular liver disease or cirrhosis;
2. Presence of liver disease with other cause (autoimmune, metabolic, medication induced);
3. BMI <25 kg/m^2;
4. Alcohol use >30 g/day;
5. Type 1 diabetes;
6. 6. History of major bariatric surgery (not including balloon / sleeve gastrectomy);
7. Weight loss or gain of 5kg or more in the past 6 months or >10% change in bodyweight in the past 12 months;
8. Contraindication for MRI;
9. Inadequate venous access;
10. Lactating/breastfeeding/pregnant at Screening or Baseline;
11. HIV antibody positive, hepatitis B surface antigen positive (HBsAg) or Hepatitis C virus (HCV)-RNA positive;
12. Receiving an elemental diet or parenteral nutrition;
13. Concurrent conditions

    * Inflammatory bowel disease;
    * Unstable angina, myocardial infarction, transient ischemic events, or stroke within 24 weeks of Screening;
    * Ongoing infectious, ongoing multi-systemic immune-mediated and/or concurrent or past malignant disease;
    * Any other concurrent condition which, in the opinion of the investigator, could impact adversely on the subject participating or on the interpretation of the study data;
14. Concurrent medications including:

    * anti-NASH therapy(s) taken for more than 10 continuous days in the last 3 months. These include S-adenosyl methionine (SAM-e), betaine, milk thistle, probiotic supplements (other than yoghurt), vitamin E and gemfibrozil.

      * NB: If vitamin E or gemfibrozil are used, the dose must be stable and liver biopsy confirming diagnosis of NASH subsequent to commencing treatment; commencing treatment;
      * Wash out for any of the anti-NASH therapies is as follows: under 10 days no washout required, more than 10 days and up to 3 months treatment requires 6 weeks washout. Any treatment of over 3 months would require to re-biopsy to ensure histological eligibility
    * thiazolidinediones (glitazones), dipeptidyl peptidase 4 inhibitors (gliptins) or glucagon-like peptide-1 analogs in the last 6 months. If treatment commenced and is stable for more than 6 month prior to the determinant biopsy and the dose is still stable at time of study entry, subjects will be eligible for recruitment.
    * Allowable anti-diabetic treatment includes metformin and/or sulfonylureas administered at constant dose for at least 2 months prior to study entry.
    * Subjects treated with Insulin are eligible if clinically stable on insulin treatment (i.e. no recurrent acute hypo-/hyperglycemic episodes diagnosed clinically and by Glucose serum levels of <50 mg/dL and >200 mg/dL respectively) for at least 2 months prior to study entry.
    * immune modulatory agents including

      * In the last 3 months:
      * systemic steroids for more than 7 days.
      * daily treatment with multiple non-steroidal anti-inflammatory drugs (such as aspirin >100mg/day, ibuprofen, naproxen, meloxicam, celecoxib) for more than 1 month within 3 months prior to study entry;
      * In the last 12 months:
      * azathioprine, 6-mercaptopurine, methotrexate, cyclosporin, anti-TNFα therapies (infliximab, adalimumab, etanercept) or anti-integrin therapies (namixilab) ;
    * more than 10 consecutive days oral or parenteral antibiotics within 4 weeks prior to study entry (Note: such subjects would not be included in the stool and PBMC analysis).
    * variable dose of antilipidemic agents (3-hydroxy-3-methyl-glutaryl (HMG)-Co-A reductase inhibitors - "statins") in the 3 months prior to study entry.
15. The following laboratory abnormalities:

    * Neutrophil count ≤1.0 x 10^9/L
    * Platelets <100 x 10^9/L
    * Hemoglobin <10 g/dL
    * Albumin <3.5 g/dL
    * International Normalized Ratio (INR) >1.5
    * Total bilirubin >1.5 x upper limit of reference range (unless Gilbert's syndrome or extrahepatic source as denoted by increased indirect bilirubin fraction)
    * Either creatinine clearance ≤60 mL/minute calculated by Cockroft Gault or creatinine >1.5x upper limit of reference range.
16. Known substance abuse, including inhaled or injected drugs in the year prior to Screening.
17. Cow milk allergy, lactose intolerance or any known or suspected hypersensitivity to study products.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2014-12; Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Peres, Study Director — Immuron Ltd.
Locations (25):
- United States (17):
  - eStudySite, Chula Vista, California
  - University of California San Diego, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - University of Florida Hepatology Research at CTRB, Gainesville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Kansas City Research Institute, Kansas City, Missouri
  - Duke Liver Centre, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Baylor St Lukes Medical Centre, Houston, Texas
  - Brooke Army Medical Centre, Houston, Texas
  - Pinnacle Clinical Research, Live Oak, Texas
  - University of Virginia Medical Centre, Charlottesville, Virginia
  - Mary Immaculate Hospital, Newport News, Virginia
  - Bon Secours St Marys Hospital, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Medical Centre, Seattle, Washington
- Australia (6):
  - The Nepean Hospital, Penrith, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - The Alfred Hospital, Prahran, Victoria
- Israel (2):
  - Hadassah Medical Centre, Jerusalem
  - Sourasky Medical Center (Ichilov), Tel Aviv

REFERENCES:
- [Derived] Nedrud MA, Chaudhry M, Middleton MS, Moylan CA, Lerebours R, Luo S, Farjat A, Guy C, Loomba R, Abdelmalek MF, Sirlin CB, Bashir MR. MRI Quantification of Placebo Effect in Nonalcoholic Steatohepatitis Clinical Trials. Radiology. 2023 Mar;306(3):e220743. doi: 10.1148/radiol.220743. Epub 2022 Nov 1. PMID 36318027
- [Derived] Jin L, Sun Y, Li Y, Zhang H, Yu W, Li Y, Xin Y, Alsareii SA, Wang Q, Zhang D. A synthetic peptide AWRK6 ameliorates metabolic associated fatty liver disease: involvement of lipid and glucose homeostasis. Peptides. 2021 Sep;143:170597. doi: 10.1016/j.peptides.2021.170597. Epub 2021 Jun 10. PMID 34118361

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Started | 43 | 46 | 44
Completed | 32 | 39 | 41
Not Completed | 11 | 7 | 3
Not completed — Adverse Event | 2 | 2 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Non compliance | 3 | 1 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — TBC | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C | Total
Number analyzed (Participants) | 43 | 46 | 44 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (11.9) | 50.2 (13.7) | 50.2 (11.1) | 50.59 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 20 | 70
  Male | 20 | 19 | 24 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 6 | 1 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 0 | 1
  White | 30 | 40 | 34 | 104
  More than one race | 2 | 2 | 2 | 6
  Unknown or Not Reported | 5 | 2 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 34 | 32 | 34 | 100
  Israel | 1 | 6 | 5 | 12
  Australia | 8 | 8 | 5 | 21
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.97 (5.439) | 34.12 (5.802) | 34.54 (5.678) | 34.21 (5.653)
HbA1c [Mean (Standard Deviation); unit: %] | 6.14 (0.765) | 6.16 (0.999) | 6.12 (0.916) | 6.141 (0.896)
Hepatic Fat [Mean (Standard Deviation); unit: %] | 19.64 (9.237) | 19.11 (8.166) | 18.39 (7.067) | 19.04 (8.219)

OUTCOME MEASURES:

1. Primary Outcome: Safety Outcome Measure
Description: Incidence of adverse events per arm/group
Time Frame: 24 Weeks
Population: Number of treatment emerged AEs per arm/group
Measure: Number; unit: AEs
Groups:
- IMM-124E, 600 mg: IMM-124E, 600 mg three times daily, orally plus matching placebo 24 weeks of treatment
- IMM-124E, 1200 mg: IMM-124E, 1200 mg three times daily, orally 24 weeks of treatment
- Matching Placebo: Matching placebo, three times daily, orally 24 weeks of treatment
Arm/Group | IMM-124E, 600 mg | IMM-124E, 1200 mg | Matching Placebo
Number analyzed (Participants) | 43 | 46 | 44
AEs | 185 | 207 | 155

2. Primary Outcome: Percentage Fat Content of the Liver
Description: Mean change from Baseline in Percentage Fat Content of the Liver measured by Magnetic Resonance Imaging (MRI) at Week 24
Time Frame: baseline and 24 weeks
Population: The analysis population includes subjects with both baseline MRI and week 24 MRI.
Measure: Mean (Standard Deviation); unit: percentage of hepatic fat fraction
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 35 | 40 | 41
percentage of hepatic fat fraction | -1.55 (0.903) | -0.90 (0.818) | -1.85 (0.810)

3. Primary Outcome: Adverse Events
Description: Number of patients with treatment-related adverse events
Time Frame: 24 weeks
Population: Number of patients with any treatment-related AE
Measure: Count of Participants; unit: Participants
Arm/Group | IMM-124E, 600 mg | IMM-124E, 1200 mg | Matching Placebo
Number analyzed (Participants) | 43 | 46 | 44
Participants | 17 | 14 | 13

4. Primary Outcome: Severity of Adverse Events
Description: Number of grade 3-5 adverse events
Time Frame: 24 weeks
Population: Number of grade 3-5 AEs
Measure: Number; unit: events
Arm/Group | IMM-124E, 600 mg | IMM-124E, 1200 mg | Matching Placebo
Number analyzed (Participants) | 43 | 46 | 44
events | 12 | 10 | 7

5. Secondary Outcome: Systolic Blood Pressure
Description: Mean change in Systolic Blood Pressure
Time Frame: baseline and 24 weeks
Population: The analysis population include subjects with data of both baseline and week 24
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 41
mmHg | 6.1 (16.19) | 2.0 (12.73) | 0.2 (14.75)

6. Secondary Outcome: Pulse Rate
Description: Mean change in Pulse Rate from baseline to week 24
Time Frame: baseline and 24 weeks
Population: The analysis population include subjects with Pulse Rate data of both baseline and week 24
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 41
beats/minute | -0.8 (10.91) | -1.9 (9.29) | 2.1 (10.00)

7. Secondary Outcome: Diastolic Blood Pressure
Description: Change in Diastolic Blood Pressure
Time Frame: baseline and 24 weeks
Population: The analysis population include subjects with data of both baseline and week 24
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 41
mmHg | 0.6 (11.17) | -0.5 (6.40) | -0.3 (8.37)

8. Secondary Outcome: Respiratory Rate
Description: Mean change in Respiratory Rate from baseline to week 24
Time Frame: baseline and 24 weeks
Population: The analysis population includes subjects with both respiratory rate data at baseline and week 24
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 41
breaths/minute | -0.2 (1.63) | -0.3 (1.68) | 0.1 (2.08)

9. Secondary Outcome: Serum Alanine Aminotransaminase (ALT)
Description: Mean change from Baseline in Serum Alanine Aminotransaminase (ALT) at Week 24
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
IU/L | -14.4 (4.95) | -10.7 (4.55) | -10.3 (4.49)

10. Secondary Outcome: Peak Serum Concentration (Cmax)
Description: Peak serum concentration (Cmax) of IMM-124E
Time Frame: 0, 4, 12 and 24 Weeks
Population: The investigational product is orally active and not systemically absorbed into the blood stream. This analysis purpose was to confirm this claim and show there is no absorption to blood stream.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
ng/mL | 0 (0) | 0 (0) | 0 (0)

11. Secondary Outcome: Minimum Serum Concentration (Cmin)
Description: Minimum serum concentration (Cmin) of IMM-124E
Time Frame: 0, 4, 12 and 24 Weeks
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
ng/mL | 0 (0) | 0 (0) | 0 (0)

12. Secondary Outcome: Area Under the Concentration Time Curve (AUC)
Description: Area Under the Concentration Time Curve (AUC) of IMM-124E. Time points at which data were collected: baseline pre-dose, week 4, week 12 and week 24.
Time Frame: 0, 4, 12 and 24 Weeks
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
ng/mL | 0 (0) | 0 (0) | 0 (0)

13. Secondary Outcome: Elimination Half Life (T1/2)
Description: Elimination Half Life (T1/2) of IMM-124E
Time Frame: 0, 4, 12 and 24 Weeks
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
seconds | 0 (0) | 0 (0) | 0 (0)

14. Secondary Outcome: Body Mass Index (BMI)
Description: Change from Baseline of Body Mass Index (BMI) at 24 weeks
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
kg/m^2 | 0.20 (1.024) | -0.33 (1.701) | 0.09 (1.350)

15. Secondary Outcome: Waist Circumference
Description: Change from Baseline of Waist Circumference at 24 weeks
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 21 | 33 | 29
cm | -1.20 (4.353) | -0.35 (5.969) | -0.92 (6.090)

16. Secondary Outcome: Waist:Hip Ratio
Description: Change from Baseline of Waist:Hip Ratio at 24 weeks
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 21 | 33 | 29
ratio | -0.02 (0.051) | 0.01 (0.063) | 0.01 (0.079)

17. Secondary Outcome: Hemoglobin (HB)A1C
Description: Change from Baseline of Hemoglobin(HB)A1C at 24 weeks
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 36 | 39
percentage | 1.0 (0.88) | 0.1 (0.84) | 0.2 (0.81)

18. Secondary Outcome: Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Description: Change from Baseline of Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at 24 weeks
Time Frame: baseline and 24 Weeks
Population: HOMA-IR is calculated according to the formula: fasting insulin (mU/mL) x fasting glucose (mmol/L)/22.5
Measure: Mean (Standard Deviation); unit: no unit
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 30 | 36 | 35
no unit | 2.098 (2.3374) | 0.057 (2.1340) | 0.655 (2.1648)

19. Secondary Outcome: Total Cholesterol
Description: Change from Baseline of Total Cholesterol at 24 weeks
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
mmol/l | -0.1 (0.11) | 0.0 (0.10) | 0.0 (0.10)

20. Secondary Outcome: Triglycerides
Description: Change from Baseline of Triglycerides at 24 weeks
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
mmol/l | -0.7 (1.25) | -0.3 (1.15) | -0.4 (1.14)

21. Secondary Outcome: Low Density Lipoprotein (LDL)
Description: Change from Baseline of Low Density Lipoprotein (LDL) at 24 weeks
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 30 | 37 | 37
mmol/l | -0.1 (0.09) | 0.1 (0.08) | 0.0 (0.08)

22. Secondary Outcome: High Density Lipoprotein (HDL)
Description: Change from Baseline of High Density Lipoprotein (HDL) at 24 weeks
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
mmol/l | 0.0 (0.03) | 0.0 (0.02) | 0.1 (0.02)

23. Secondary Outcome: Serum Alanine Aminotransaminase (ALT)
Description: Mean change from Baseline of serum ALT
Time Frame: baseline to 24 weeks
Population: assessed at 0, 4, 8, 12, 16, 20 and 24 Weeks, change from baseline to week 24 reported
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
IU/L | -14.4 (4.95) | -10.7 (4.55) | -10.3 (4.49)

24. Secondary Outcome: Serum Aspartate Aminotransaminase (AST)
Description: Mean change from Baseline of Serum AST
Time Frame: baseline to 24 Weeks
Population: assessed at 0, 4, 8, 12, 16, 20 and 24 Weeks, change from baseline to week 24 reported
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
IU/L | -7.8 (3.32) | -7.4 (3.05) | -7.5 (3.01)

25. Secondary Outcome: Bilirubin
Description: Mean change from Baseline of Bilirubin
Time Frame: baseline to 24 Weeks
Population: assessed at 0, 4, 8, 12, 16, 20 and 24 Weeks, change from baseline to week 24 reported
Measure: Mean (Standard Deviation); unit: umol/l
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
umol/l | -1.0 (3.56) | -1.0 (0.54) | 0.3 (0.53)

26. Secondary Outcome: Albumin
Description: Mean change from Baseline of Albumin
Time Frame: baseline to 24 Weeks
Population: assessed at 0, 4, 8, 12, 16, 20 and 24 Weeks, change from baseline to week 24 reported
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
g/dL | -0.8 (0.35) | -0.2 (0.32) | 0.3 (0.32)

27. Secondary Outcome: Gamma Glutamyl Transpeptidase (GGT)
Description: Mean change from Baseline of Gamma Glutamyl Transpeptidase (GGT)
Time Frame: baseline to 24 Weeks
Population: assessed at 0, 4, 8, 12, 16, 20 and 24 Weeks, change from baseline to week 24 reported
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
U/L | -7.1 (5.03) | -9.7 (4.62) | -5.7 (4.56)

28. Secondary Outcome: Serum Alanine Aminotransaminase (ALT)
Description: Number of patients with ALT within the normal reference range at Week 24 (defined a <19 IU/L for women and <30 IU/L for men)
Time Frame: 24 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 40
Participants | 3 | 4 | 2

29. Other Pre Specified Outcome: Serum Concentrations of Lipopolysaccharide (LPS)
Description: The percentage of subjects reporting at least 15% reduction in LPS, from baseline to Week 24
Time Frame: 0, 4, 12 and 24 Weeks
Population: excluding subjects with < 250 LPS at baseline (comparing 1200mg IMP group to Placebo group). PP population, excluding outliers sites. this Outcome Measure was pre-specified to be assessed in the 1200mg and Placebo Arms/Groups *only*
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 0 | 28 | 29
Participants |  | 18 | 10

30. Other Pre Specified Outcome: Regulatory T Cells (FoxP3+ CD25-CD4+) in Peripheral Blood Mononuclear Cells
Description: Change in percent of FoxP3+ CD25-CD4+ cells in Peripheral Blood Mononuclear Cells
Time Frame: 0 and 24 Weeks
Population: Sub group population with PBMC FACS data, selected sites only.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | IMM-124E, 600 mg | IMM-124E, 1200 mg | Matching Placebo
Number analyzed (Participants) | 1 | 8 | 3
percentage of cells | NA (NA) — only 1 participant's data analyzed in 600mg arm. | 0.46 (0.26) | 14.59 (14.58)

31. Other Pre Specified Outcome: Gut Microbiome From Fecal Samples
Description: Number of participants with measurable differences in gut microbiome constituents post-treatment
Time Frame: 0, 4, 12 and 24 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 4 | 12 | 5
Participants | 0 | 0 | 0

32. Other Pre Specified Outcome: Serum Concentrations of LPS
Description: Serum Concentrations of Lipopolysaccharide (LPS) (ng/mL) levels and change from Baseline
Time Frame: baseline to 24 Weeks
Population: assessed at 0, 4, 12 and 24 Weeks, change from baseline to week 24 reported
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 33 | 39 | 35
ng/mL | -130.763 (188.153) | 78.488 (173.029) | 414.912 (182.632)

33. Other Pre Specified Outcome: Serum Concentrations of C-Reactive Protein (CRP)
Description: Mean Serum Concentrations of C-Reactive Protein (CRP) at week 24
Time Frame: baseline to 24 Weeks
Population: assessed at 0, 4, 12 and 24 Weeks, change from baseline to week 24 reported
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 35 | 40 | 41
mg/L | 0.711 (0.68) | 1.129 (1.637) | 1.364 (2.317)

34. Other Pre Specified Outcome: Serum Concentrations of CK-18 Fragments
Description: The proportion of subjects with significant reduction of CK-18 (≥ 15%) between IMP 1200mg group to placebo.
Time Frame: baseline to 24 weeks
Population: FAS population, excluding outlier sites. this Outcome Measure was pre-specified to be assessed in the 1200mg and Placebo Arms/Groups *only*
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 0 | 36 | 33
Participants |  | 14 | 6

35. Other Pre Specified Outcome: Serum Concentrations of Human Adiponectin
Description: Change from Run-in to Post-treatment in serum concentration of human Adiponectin.
Time Frame: 0 to 24 Weeks
Population: ITT population. Run-in = mean of screening and baseline values. assessed at 0, 4, 12 and 24 Weeks, change from baseline to week 24 reported
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 38 | 43 | 37
pg/mL | 107560.15 (1082735.0) | 208185.48 (1115352.8) | 1082735.0 (1900710.5)

36. Other Pre Specified Outcome: Serum Concentrations of Cytokine IL-6
Description: Mean Change from baseline to week 24 of serum concentration of cytokine IL-6
Time Frame: 24 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 36 | 41 | 39
pg/mL | 0.1234 (0.90505) | 0.1031 (1.63948) | 0.4117 (1.50248)

37. Other Pre Specified Outcome: Serum Concentration of Cytokine IL-12p70
Description: Mean change from baseline to week 24 of Serum concentration of Cytokine IL-12p70
Time Frame: 24 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 36 | 41 | 39
pg/mL | 0.0494 (1.00060) | 0.3274 (2.76062) | 0.0579 (1.35852)

38. Other Pre Specified Outcome: Serum Concentration of Interferon Gamma (IFN-γ)
Description: Mean Change from baseline to week 24 of serum concentration of IFN-gamma
Time Frame: 24 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 36 | 41 | 39
pg/mL | 0.9523 (6.25581) | 0.8058 (6.59164) | 1.4514 (7.56336)

39. Other Pre Specified Outcome: Serum Concentration of Tumor Necrosis Factor Alpha (TNF-α)
Description: Mean Change from baseline to week 24 of serum concentration of TNF-α
Time Frame: 24 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 36 | 41 | 39
pg/mL | -0.1691 (1.68068) | -0.5082 (1.59892) | -0.3877 (2.16469)

40. Other Pre Specified Outcome: Serum Concentration of Glucagon-like Peptide-1 (GLP-1)
Description: Mean Change from baseline to week 24 of serum concentration of GLP-1
Time Frame: 24 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: pM
Arm/Group | Treatment Arm A | Treatment Arm B | Treatment Arm C
Number analyzed (Participants) | 37 | 41 | 39
pM | 1.6457 (15.79917) | -1.5310 (13.07262) | 3.4820 (33.36977)

41. Other Pre Specified Outcome: Regulatory T Cells (FoxP3+CD25-CD8+) in Peripheral Blood Mononuclear Cells
Description: Change in percent of FoxP3+CD25-CD8+ cells in Peripheral Blood Mononuclear Cells
Time Frame: 0 and 24 Weeks
Population: Sub group population with PBMC FACS data, selected sites only.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | IMM-124E, 600 mg | IMM-124E, 1200 mg | Matching Placebo
Number analyzed (Participants) | 1 | 8 | 3
percentage of cells | NA (NA) — only 1 participant's data analyzed in 600mg arm. | -0.01 (0.33) | 12.52 (12.32)

ADVERSE EVENTS:
Time Frame: 28 weeks after participant received first dose
Description: The adverse event information collected in the clinical study is collected based on the adverse event definition of ''Results Data Element Definitions for Adverse Events''.
  The adverse events data was collected based on physician's assessments, laboratory assessments, subjects reporting and questionnaires.
Arm/Group | IMM-124E, 600 mg | IMM-124E, 1200 mg | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/46 | 1/44
Serious Adverse Events (participants affected / at risk) | 1/43 | 2/46 | 3/44
Other Adverse Events (participants affected / at risk) | 39/43 | 41/46 | 38/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMM-124E, 600 mg (N=43) | IMM-124E, 1200 mg (N=46) | Matching Placebo (N=44)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Psychiatric hospitalisation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMM-124E, 600 mg (N=43) | IMM-124E, 1200 mg (N=46) | Matching Placebo (N=44)
Nausea (Gastrointestinal disorders) | 8 (10) | 15 (16) | 11 (16)
Fatigue (General disorders) | 8 (10) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 11 (16) | 8 (17) | 8 (10)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 6 (6) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (11) | 6 (8) | 9 (10) — lower and/or upper
Constipation (Gastrointestinal disorders) | 4 (6) | 7 (8) | 4 (4)
Flatulence (Gastrointestinal disorders) | 5 (5) | 5 (6) | 4 (5)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (4) | 5 (7)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 2 (5)
Sinusitis (Infections and infestations) | 2 (3) | 3 (4) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (6) | 5 (5)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (4)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 5 (7) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT02316717/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT02316717/SAP_001.pdf